CLINICAL TRIAL: NCT04919902
Title: Prague Registry of Electric Cardioversion for Supraventricular Arrhythmias
Brief Title: Prague Registry of Electric Cardioversion
Acronym: PRAGUE-ECV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Marek Sramko, Head of the Department of Acute Cardiology, Institute for Clinical and Experimental Medicine
Other Study IDs: EKV2020
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Atrial Arrhythmia; Atrial Tachycardia
Keywords: Anticoagulants; Anticoagulation; Cardioversion; NOAC; DOAC
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Electric Countershock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Electric cardioversion: Patients who underwent elective cardioversion for atrial arrhythmia
  Interventions: Procedure: Electric cardioversion

INTERVENTIONS:
Procedure: Electric cardioversion — Electric cardioversion in short sedation according to established clinical practice and indications

SUMMARY:
This single-center observational registry follows contemporary efficacy and short-term complications of elective electric cardioversion.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive out-patients undergoing electric cardioversion for atrial fibrillation, atrial tachycardia, or typical atrial flutter

Exclusion Criteria:

* Unstable patients with acute conditions requiring unplanned hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodynamically stable patients scheduled for ambulatory electric cardioversion for atrial arrhythmias based on established clinical indications.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Acute major complications | Within 24 hours from the procedure
  Major thromboembolic events or events related to cardioversion requiring unplanned hospitalisation (bleeding, severe bradycardia, anesthesia-related complications, heart failure etc)
Subacute major complications | 24 hours to 30 days after the procedure
  Major thromboembolic events or events related to cardioversion requiring unplanned hospitalisation (bleeding, severe bradycardia, anesthesia-related complications, acute heart failure etc), evaluated by structured phone call.

SECONDARY OUTCOMES:
Acute minor complications | Within 24 hours from the procedure
  Minor procedure-related complications not requiring acute hospitalisation (asymptomatic bradycardia, post-anesthesia spasms)
Acute efficacy | Within 2 hours from the procedure
  Presence of sinus rhythm on continous ECG (5-lead) monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided